CLINICAL TRIAL: NCT02094846
Title: Evaluation of the Effect of an Intervention Based on Cell Phones on Glycemic Control in Adults With Type 2 Diabetes Mellitus
Brief Title: Evaluation of an Intervention Based on Cell Phones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Salud Publica, Mexico (Other)
Responsible Party: Principal Investigator, Mario Efraín Flores Aldana, Jefe del Departamento de Epidemiología Nutricional. Centro de Investigación en Nutrición y Salud, Instituto Nacional de Salud Publica, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Evaluation with cell phones
Record Dates: First submitted 2014-03-04; First posted 2014-03-24 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Cellular phones; Type 2 diabetes; Glycated hemoglobin; glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Voice messages (Active Comparator): This group receive voice messages to reinforce given information about diet, physical activity, glycemic index
  Interventions: Behavioral: Voice messages
- Messages (Placebo Comparator): This group received voice messages with fun facts.

INTERVENTIONS:
Behavioral: Voice messages — Voice messages reinforced with self-efficacy
  Arms: Voice messages

SUMMARY:
The aim of the study was to assess the effect of an individualized intervention based on cell phones to improve glycemic control in patients with type 2 diabetes attending Epidemiology Research Unit in Cuernavaca, Morelos. Mexico

DETAILED DESCRIPTION:
In this study before randomization, the participants received workshops on diet, physical activity, glycemic index of foods.

Bandura´s theoretical model was used in the voice messages sent to the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus > 10 years
* Glycated hemoglobin >7%

Exclusion Criteria:

* Take insulin regularly
* Pregnant woman
* Woman who expected to be pregnant the next 6 months
* 24 hrs creatinine < 30 ml/minute

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin | Basal and 3 months
  Glycated hemoglobin is obtained from a blood sample at the beginning of the study and 3 months later.

SECONDARY OUTCOMES:
Low Density Lipoprotein | Basal and 3 months
  Low Density Lipoprotein is obtained from a blood sample at the beginning of the study and 3 months later.
High Density Lipoprotein | Basal and 3 months
  High Density Lipoprotein is obtained from a blood sample at the beginning of the study and 3 months later.
Cholesterol | Basal and 3 months
  Cholesterol is obtained from a blood sample at the beginning of the study and 3 months later.
Self-efficacy | Basal and 3 months
  Self-efficacy questionnaire is divided into a diet´s self-efficacy questionnaire and physical activity´s self-efficacy questionnaire.
  People can obtained "low self-efficacy" status or "high self-efficacy" status
Physical activity | Basal and 3 months
  A triaxial accelerometer was used, colocated on the hip and the participants were supposed to use it 7 days for a minimal of 10 hours per day

CONTACTS AND LOCATIONS:
Overall Officials: Mario E Flores Aldanda, PhD, Principal Investigator — Instituto Nacional de Salud Pública
Locations (1):
- Unidad de Investigación en Epidemiología y Servicios de Salud del Instituto Mexicano del Seguro Social, Cuernavaca, Morelos, Mexico

REFERENCES:
- [Background] Oh JA, Kim HS, Yoon KH, Choi ES. A telephone-delivered intervention to improve glycemic control in type 2 diabetic patients. Yonsei Med J. 2003 Feb;44(1):1-8. doi: 10.3349/ymj.2003.44.1.1. PMID 12619168
- [Background] Liang X, Wang Q, Yang X, Cao J, Chen J, Mo X, Huang J, Wang L, Gu D. Effect of mobile phone intervention for diabetes on glycaemic control: a meta-analysis. Diabet Med. 2011 Apr;28(4):455-63. doi: 10.1111/j.1464-5491.2010.03180.x. PMID 21392066
- [Background] Cole-Lewis H, Kershaw T. Text messaging as a tool for behavior change in disease prevention and management. Epidemiol Rev. 2010;32(1):56-69. doi: 10.1093/epirev/mxq004. Epub 2010 Mar 30. PMID 20354039
- See also: Effectiveness of mobile and internet intervention in patients with obese type 2 diabetes — http://www.ncbi.nlm.nih.gov/pubmed/17881285